CLINICAL TRIAL: NCT05518084
Title: Evaluating the Safety and Tolerability of the Liponovo Tissue Product in Healthy Volunteers
Brief Title: Safety of Cell-free Adipose Tissue Product in Healthy Volunteers
Acronym: SAFETY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linio Biotech Oy (Industry)
Collaborators: Clinius Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-001
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Safety Issues

STUDY DESIGN:
Intervention Model Description: Participants are not randomized into different arms. Instead, the side (left or right forearm) receiving the investigational product vs. placebo is randomized for each participant.
Masking Description: Participants and investigators are blinded to which arm receives placebo vs. investigational product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liponovo tissue product and Ringer Acetat injections (Experimental): Investigational products (Liponovo tissue product and Ringer Acetat) are injected into the dorsal forearm, superficial part of the subcutis.
  Interventions: Other: Liponovo tissue product

INTERVENTIONS:
Other: Liponovo tissue product — Investigational products (Liponovo tissue product and Ringer Acetat) are injected into the dorsal forearm, superficial part of the subcutis. The single injection and a 23G/30mm needle are used. The amount of the injected investiogational products is 4,5 ml for both dorsal forearms (together 4,5ml x2 = 9ml / test subject). The product is always injected in the proximal third of the forearm, into a standardized a quarter circle with a radius of 30mm. Both injections are performed with covered syringe to ensure the double-blinding. After the injection, test subjects get a cold on the injection sites to reduce the bruising.

SUMMARY:
The study is a randomized, double blinded, bilaterally controlled trial.The aim is to evaluate the short- and mid term safety of cell-free adipose tissue product. The safety of the tissue product is to be studied in 40 healthy volunteers. Cell-free tissue product is injected into superficial part of the subcutis with one injection to standardized area. The volume of the injection is 4,5 ml. As the control method, the same size area is injected with plain Ringer-Acetat solution. The adverse events and serious adverse events are monitored in doctor visits, phone calls and e-diary.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 years or more)
* Healthy skin in the studied area (dorsal forearm, proximal third)
* Able and willing to give informed consent
* Reasonably accessible to the study clinic and compliant to follow-up visits

Exclusion Criteria:

* known allergy to any of the preparations used in the study (Liponovo tissue product and Ringer-Acetat) or earlier/known anaphylaxis reaction for any allergen
* hematologic or other bleeding disorder
* use of antitrombotic/ anticoagulation medicine
* autoimmune disease
* immunosupressive disease or medication
* cancer or neoplastic disease
* connective tissue disease
* diabetes type 1 or 2 or other metabolic diseases
* smoking
* pregnancy or nursing
* sunbathing during last 7 days
* a skin disease that is or has been symptomatic in the studied area
* test subjects with previous fat or hyaluronic acid filling under the same area
* those who withhold consent
* Use of following medications:
* Histamine receptor-blockers <7 days before study initiation
* Topical corticosteroids in test area <7 days before study initiation
* Topical calsineurin inhibitors <7days before study initiation
* Longterm (>10days before study initiation) systemic prednisolon >10mg/d
* Omalitsumabi < 4weeks before study initiation
* Doksepin < 7 days before study initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Acute local reactions 20 minutes after injection | Day 0
  Examination and structured interview 20 minutes after injection by the investigator
Acute and mid-term adverse events, incl severe adverse events | Day 0-7, Day 30, and Day 60
  E-dairy filled out by the participants
Acute and mid-term adverse events, incl severe adverse events | Day 90
  Evaluation and structured interviews by the investigator
Acute and mid-term adverse events, incl severe adverse events | Day 7 and Day 9
  Structured telephone interview by study nurse
Delayed allergic reactions | Day 0-7, Day 30, and Day 60
  Participant's e-dairy
Delayed allergic reactions | Day 2, and Day 7
  Telephone interviews by the study nurse

CONTACTS AND LOCATIONS:
Locations (1):
- Terveystalo, Ruoholahti, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No